CLINICAL TRIAL: NCT04053920
Title: Resistance Exercise Training at Different Intensities in Healthy and Frail Older People: A Feasibility Study
Brief Title: Resistance Exercise Training at Different Intensities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Stuart Gray, Senior Lecturer in Exercise and Metabolic Health, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 236559
Record Dates: First submitted 2019-08-09; First posted 2019-08-13 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Sarcopenia; Frailty; Aging
MeSH Terms: conditions — Sarcopenia; Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low load (Experimental): Training at 30-40% one-repetition maximum (1RM)
  Interventions: Behavioral: Low Load Resistance exercise
- High load (Experimental): Training at 65-75% one-repetition maximum (1RM)
  Interventions: Behavioral: High Load Resistance exercise

INTERVENTIONS:
Behavioral: Low Load Resistance exercise — leg extension, leg press, leg curl and calf press
  Arms: Low load
Behavioral: High Load Resistance exercise — leg extension, leg press, leg curl and calf press
  Arms: High load

SUMMARY:
The aim of the current study, therefore, is to determine the feasibility of recruitment and adherence to resistance exercise training interventions performed at low and high loads, to volitional muscular failure, in a trial population that includes both healthy and frail older people.

ELIGIBILITY:
Inclusion Criteria:

* Over age of 65 years

Exclusion Criteria:

* Current participation in an exercise programme
* Exercise deemed unsafe by clinical team

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
Muscle strength | Change from baseline to 8 weeks
  Knee extensor maximal torque during an isometric MVC

SECONDARY OUTCOMES:
Vastus lateralis muscle thickness | Change from baseline to 8 weeks
  Measured via ultrasound
Muscle strength | Change from baseline to 8 weeks
  Knee flexor maximal torque during an isometric MVC
One-repetition maximum | Change from baseline to 8 weeks
  leg extension, leg curl, leg press and calf press
Biomechanics during walking and stair climbing | Change from baseline to 8 weeks
  Motion analysis
Short performance physical battery test | Change from baseline to 8 weeks
  SPPB - balance, walking pace and chair rise
Quality of life measure | Change from baseline to 8 weeks
  EQ-5D-5L questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Gray, Principal Investigator — University of Glasgow
Locations (1):
- GRI Clinical Research Facility, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No